CLINICAL TRIAL: NCT01662570
Title: Beverage Choice and Lifestyle Modification in Overweight Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 807775; R21DK079075 (NIH)
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2011-11

CONDITIONS: Obesity
Keywords: Pediatric Obesity; Child Overweight
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beverage Choice Lifestyle Modification (Active Comparator): The family-based BCLM intervention trained children and parents in self monitoring of sugar sweetened beverage intake and goal-setting, incorporated feedback and reinforcement, and provided water bottles and water filters to promote a reduction in sugar sweetened beverages and overall energy intake.
  Interventions: Behavioral: Beverage Choice and Lifestyle Modification
- Nutrition Education (NE) (Other): This treatment for parents and children addressed a variety of topics in nutrition including benefits of fruits and vegetables, the food pyramid, vitamins, benefits of eating a variety of foods, and healthy beverage selections. No behavioral change training component was included.
  Interventions: Other: Nutrition Education (NE)

INTERVENTIONS:
Behavioral: Beverage Choice and Lifestyle Modification — The family-based BCLM intervention trained children and parents in self monitoring of sugar sweetened beverage intake and goal-setting, incorporated feedback and reinforcement, and provided water bottles and water filters to promote a reduction in sugar sweetened beverages and overall energy intake. 16 sessions were provided over a 6-month period.
  Arms: Beverage Choice Lifestyle Modification
Other: Nutrition Education (NE) — This treatment for parents and children addressed a variety of topics in nutrition including benefits of fruits and vegetables, the food pyramid, vitamins, benefits of eating a variety of foods, and healthy beverage selections. No behavioral change training component was included. 16 sessions over 24 weeks was provided.
  Other Names: NE
  Arms: Nutrition Education (NE)

SUMMARY:
The rise in childhood overweightness and concomitant increase in chronic disease risk warrants exploration into the effectiveness of interventions targeting the eating and activity habits of overweight youth. This research study developed and tested a "Beverage Choice and Lifestyle Modification" (BCLM) intervention for 4 to 8 year old children who are at-risk for being overweight or are overweight and who consume large amounts of sugar sweetened beverages and juice. The overall study objectives were to test the acceptability and effectiveness of the BCLM intervention for improving the weight status, energy (kcal) intake, beverage selections and beverage preferences of children in targeted age and BMI group. The investigators hypothesized that those children randomized to the BCLM group will show greater improvements in weight and Body Mass Index (BMI) status, beverage choices,and energy intake than those assigned to our Nutrition Education (NE) group.

ELIGIBILITY:
Inclusion Criteria:

* Ages 4-8 years old
* BMI≥85th percentile (based on age and sex)
* consumes large (≥16 oz.day) sugar sweetened beverages

Exclusion Criteria:

* Child has a serious medical condition
* Signs of elevated psychopathology are present, as assessed by the Child Behavior Checklist (CBCL)
* Parent demonstrates elevated psychiatric problems or eating disorders
* Failure of parent or child to meet BMI criteria

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Baseline and Month 6
  Change in BMI will be measured from baseline to end of treatment (month 6).
Body Mass Index z-score (BMI-z) | Baseline and month 6
  Change in BMI-z will be measured from baseline to end of treatment (month 6).
Body Mass Index Percentile (BMI%) | Baseline and Month 6
  Change in BMI% will be measured from baseline to end of treatment (month 6).
Child percent overweight | Baseline and Month 6
  Change in child percent overweight will be measured from baseline to end of treatment (month 6).
Waist Circumference | Baseline to Month 6
  Change in waist circumference will be measured from baseline to end of treatment (month 6).
Energy (kcal) intake | Baseline to Month 6
  Change in energy intake (kcals/day) will be measured from baseline to end of treatment (month 6) using 3-day food diaries.
Sugar-sweetened beverage intake | Baseline to Month 6
  Change in sugar-sweetened beverage intake will be measured from baseline to end of treatment (month 6).
Treatment acceptance and satisfaction | Month 6
  Overall treatment acceptance and satisfaction will be measured at end of treatment.

SECONDARY OUTCOMES:
Child preferences and motivation for sugar-sweetened beverages | Baseline and Month 6
  Change in child preference and motivation for sugar-sweetened beverages will be measured from baseline to month 6 using a computerized behavioral choice task assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Myles S Faith, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States